CLINICAL TRIAL: NCT05102669
Title: Spike-specific Cellular Immune Response After COVID-19 Vaccination
Acronym: RIS-COV
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 20/09
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: COVID19; Vaccination; Immune Response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — whole blood samples and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vaccinated: COVID19 vaccinated subjects
  Interventions: Other: analysis of immunological response; Diagnostic Test: analysis of serum antibodies
- non vaccinated: COVID19 non vaccinated subjects
  Interventions: Other: analysis of immunological response

INTERVENTIONS:
Other: analysis of immunological response — collection and analysis of SARS-CoV2 Spike specific blood cells
Diagnostic Test: analysis of serum antibodies — analysis of anti-SARS-CoV2 Spike specific antibodies
  Groups: vaccinated

SUMMARY:
Aim of this study is to evaluate whether COVID-19 vaccination induces a persistent cellular immune response.

To this aim, blood samples are taken from vaccinated individuals and not immunized subjects as a control group.

Cells isolated from blood samples are tested in vitro to assess the percentage of spike-specific T and B lymphocytes 1 and 7 months after a second dose of Comirnaty vaccine.

DETAILED DESCRIPTION:
After providing written informed consent, 28 vaccinated and 25 non vaccinated subjects were included in the study. All subjects were enrolled among healthcare workers in the Research Centre of IRCCS San Raffaele Roma in Rome.

All the subjects declared that they never tested positive for COVID19. Blood and serum samples were drowned twice from vaccinated subjects: 1 and 7 months after a second dose of vaccine to evaluate T and B response to vaccine; blood was drowned once in not vaccinated subjects.

Cells were collected form peripheral blood samples, while anti-S1 IgG titre was assessed in serum.

Flow-cytometry was used to assess the percentage of circulating spike-specific T and B lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* vaccinated and non vaccinated subjects
* subjects that never tested positive for COVID19

Exclusion Criteria:

* subjects that tested positive for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IRCCS San Raffaele Roma health care workers
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
measurement of cellular response | 7 months
  evaluation of the increase of Spike-specific B and T cells percentage after COVID-19 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vitiello, PhD, Principal Investigator — IRCCS San Raffaele Roma
Locations (1):
- IRCCS San Raffaele Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided